CLINICAL TRIAL: NCT03793738
Title: Anterior Component Separation Versus Posterior Component Separation for Repair of Large Ventral Hernias: a Prospective Cohort Study
Brief Title: Anterior Component Separation Versus Posterior Component Separation for Repair of Large Ventral Hernias
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zaza Demetrashvili (Other)
Responsible Party: Sponsor-Investigator, Zaza Demetrashvili, Associate Professor, Surgery Department, Tbilisi State Medical University
Organization: Tbilisi State Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01004006344
Record Dates: First submitted 2018-12-27; First posted 2019-01-04 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Large Midline Ventral Hernia
Keywords: anterior component separation, TAR
MeSH Terms: conditions — Absent radii and thrombocytopenia

ARMS (2):
- anterior component separation (Active Comparator): The anterior component separation technique requires an extensive subcutaneous flap elevation, incision of the external oblique aponeurosis, and incision of the posterior rectus sheath.
  Interventions: Procedure: Anterior component separation
- posterior component separation (Active Comparator): The posterior component separation technique utilized the retromuscular space, accessed by incising the posterior rectus sheath and dissecting the posterior sheath between the internal oblique and transversus abdominis muscles.
  Interventions: Procedure: Posterior component separation

INTERVENTIONS:
Procedure: Anterior component separation
  Arms: anterior component separation
Procedure: Posterior component separation
  Arms: posterior component separation

SUMMARY:
This study evaluates effect of anterior component separation and posterior component separation and transversus abdominis muscle release methods for treatment of midline ventral hernias.

DETAILED DESCRIPTION:
The anterior component separation technique requires an extensive subcutaneous flap elevation, incision of the external oblique aponeurosis, and incision of the posterior rectus sheath.

The posterior component separation technique utilized the retromuscular space, accessed by incising the posterior rectus sheath and dissecting the posterior sheath between the internal oblique and transversus abdominis muscles. Transversus abdominis muscle release dissected the posterior sheath back to the transversus abdominal muscle and accessed the space between muscle and trasversalis fascia.

ELIGIBILITY:
Inclusion Criteria:

* subject has midline ventral hernia
* patient's approval to participate in the study

Exclusion Criteria:

* strangulated hernia
* patient's preference for either operative technique
* patient's refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Hernia recurrence | during 3 year after surgery
  Develop of ventral hernia recurrence

SECONDARY OUTCOMES:
Wound complications | 30 day after surgery
  Develop of wound complications (seroma, hematoma, surgical site infection)

CONTACTS AND LOCATIONS:
Overall Officials: Zaza Demetrashvili, PhD, Principal Investigator — Tbilisi State Medical University
Locations (1):
- Tbilisi State Medical University, Tbilisi, Georgia